CLINICAL TRIAL: NCT04545775
Title: KArukera Study of Ageing in Foster Families
Acronym: KASAF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Collaborators: Conseil Départemental de la Guadeloupe (Unknown)
Responsible Party: Sponsor
Other Study IDs: PAP_RIPH3_2020/01; 2020-A00620-39 (Other: ANSM)
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Geriatric Syndromes
Keywords: Older people; foster family; hospitalization; geriatric syndromes; mortality; quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Foster care for dependent older people could be a viable alternative to nursing homes. While this type of accommodation appears to be less expensive than living in a geriatric institution, few scientific studies have been able to assess its effectiveness and efficiency. In Guadeloupe, in the French West Indies, nearly 300 dependent older people are cared for by foster families. The aim of the Karukera Study of Ageing in Foster Families (KASAF) is to study the care pathways of dependent elderly people in foster care over a year. The main objective will be to obtain the annual rate of hospitalisation in this setting. The secondary objectives will be to assess hospitalisations costs, the incidence of mortality, the prevalence of geriatric syndromes, as well as the quality of life of residents and foster caregiver burnout. Ultimately, these results will be compared to a similar study in nursing homes, the KASEHPAD study (for Karukera Study of Aging in Nursing Homes).

DETAILED DESCRIPTION:
Foster care for older people is an alternative solution to nursing homes, where the resident, while still moving out of his/her own home, is taken care of within the foster family instead of a collective setting. Foster caregivers, after getting official approval and attending a 20-hour training course, usually accommodate 1 to 3 people in exchange for a monthly fee. Their mission is to ensure the well-being of their residents, and to enable them to maintain close social and family relationships. Other professionals may also provide additional nursing care if necessary. Little is known about the characteristics of foster caregivers and their residents. Epidemiological and medico-economic data on older people in foster families are essential to assess the relevance of this type of care, and several and yet unanswered questions come to mind: what is the residents' annual hospitalization rate and the associated costs? What is the prevalence of geriatric syndromes in this population, and the incidence of mortality? What is the incidence of pneumonia, the leading cause of death and emergency hospitalization in older people? What is the quality of life of the older residents and their foster caregivers? KASAF, an epidemiological cohort, aims to answer these questions. This longitudinal study will assess the health status and medical and economic data of 250 foster family residents and their foster caregivers over a year. A similar study (KASEHPAD, for Karukera Study of Aging in Nursing Homes) will be conducted simultaneously among 500 nursing home residents, as to compare these two types of care.

The main outcome is the number of hospitalizations over a year. Local PMSI (Medicalization program of the information system) hospitals databases will provide information on hospital admissions.

250 people aged 60 and older and living in foster families in Guadeloupe will be included. Data collection will be conducted using face-to-face interviews with the participants and their foster caregivers at baseline and after 6 and 12 months, and phone interviews with the foster caregivers, after 3 and 9 months. Anthropometric measures, information on general health status and care pathways (hospitalization, medical and paramedical consultations), as well as data on medical history, cognition, nutritional status, and physical frailty will also be collected. Depressive and anxiety symptoms will also be assessed along with functional abilities (mobility, instrumental activities of daily living and activities of daily living). A systematic update of vital status (death) and care pathway will be carried out at each follow-up. Additional information on the residents' living status and potential hospitalizations will be collected after 3 and 9 months. Finally, foster caregivers will be interviewed at inclusion, after 6 months and after a year to assess their own quality of life and burnout symptoms.

This study was supported by a grant from the Conseil Départemental de la Guadeloupe, Saint-Martin and Saint-Barthélemy.

ELIGIBILITY:
Inclusion Criteria:

* participant must be over 60 years old
* residents must live in a foster family in Guadeloupe, Saint-Martin or Saint-Barthelemy
* residents must benefit from the French social security
* Participant must have an identified support person
* Participant under guardianship or curatorship if accepted by the legal guardian
* Participant in a foreseeable short-term end-of-life situation if accepted by the legal representative or the support person

Exclusion Criteria:

* refusal from the resident or his legal guardian to participate in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Every elderly person living in a foster family in Guadeloupe will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-05-13 (Estimated); Study Completion 2022-11-13 (Estimated)

PRIMARY OUTCOMES:
Hospitalization rate of the participant | 12 months
  Number of hospital admissions over a year, retrieved from the local PMSI (Medicalization program of the information system) of the Hospital Center of Guadeloupe

SECONDARY OUTCOMES:
Length of hospital stays of the participant | 12 months
  Length of hospital stays expressed as number of days and nights, retrieved from the local PMSI (Medicalization program of the information system) of the Hospital Center of Guadeloupe

OTHER OUTCOMES:
Medical consultations of the participant | 12 months
  Number of consultations with a general practitioner, a medical specialist or paramedical professional will be collected.
  This information will be retrieved from the CRF using the RUD-Lite scale (Resource Utilization in Dementia questionnaire). This scale assesses the use of healthcare resources by people suffering from dementia. The foster caregiver will complete this questionnaire at inclusion and at subsequent follow-ups (T3, T6, T9 and T12).
Global cost of hospitalization of the participant | 12 months
  Global cost of hospitalization will be retrieved from the local PMSI (Medicalization program of the information system) databases after study completion
Vital status of the participant | 12 months
  Vital status (alive or deceased) will be collected at T3, T6, T9 and T12, from the foster caregiver.
Lower respiratory tract infections of the participant | 12 months
  Occurrence of lower respiratory tract infections will be collected using the RUD-lite. For the diagnosis of lower respiratory tract infections, at least two of the following must be present and a doctor must confirm the clinical evidence: Cough (starting or worsening) that may produce phlegm, specific clinical signs during auscultation; Fever. (≥38°C); Chest pain ; Rapid, shallow breathing ((≥25 per minute) ; Confusion or increased dependency.
  The foster caregiver will complete this question at inclusion and at subsequent follow-ups (T3, T6, T9 and T12).
Falls of the participant | 12 months
  Total number of falls since the last visit will be collected at T6 and T12 from the foster caregivers.
Cognition of the participant | 12 months
  The level of cognitive deterioration of the participants will be with the Mini Mental State Examination (MMSE). This 30-item scale assesses the severity of cognitive deterioration through items of orientation, learning, attention and arithmetic, memory, language, and constructive praxis.
  The scale is rated from 0 to 30, reflecting the level of cognitive impairment. The participant will complete this questionnaire at inclusion, T6 and T12.
Depressive symptoms of the participant | 12 months
  Depressive symptoms will be assessed using the CES-D (Center for Epidemiologic Studies- Depression Scale validated in French by Fuhrer & Rouillon This 20-item questionnaire assesses depressive symptomatology, including 4 items on positive affect (happiness, self-worth, confidence, enjoyment). Frequency of symptom occurrence during the past week is assessed by the participant using a 4-point Likert scale ("never", "occasionally", "quite often" and "frequently"). The score ranges from 0 to 60. The higher the score, the more significant the symptomatology. Data will be collected at inclusion, T6 and T12. For statistical analyses, the variable will be dichotomized (1 = presence of depression and 0 = absence of depression). The participant will complete this questionnaire at inclusion, T6 and T12.
Feeling of loneliness of the participant | 12 months
  Feeling of loneliness will be captured with the 14th item of the CES-D (14, 15): " I felt lonely ". The participant will complete this test at inclusion, T6 and T12
Polypharmacy of the participant | 12 months
  Total number of medications taken by participants will be collected from the foster caregiver at inclusion, T6 and T12 to assess polypharmacy.
Malnutrition of the participant | 12 months
  Malnutrition will be assessed with the short version of the Mini Nutritional Assessment (18). This questionnaire assesses nutritional status. A score under 12 indicates probable undernutrition. For the analyses, the variable will be dichotomized accordingly (1 = undernutrition; 0 = no undernutrition). The participant will complete this questionnaire at inclusion, T6 and T12.
Sarcopenia of the participant | 12 months
  The Short Physical Performance Battery (SPPB) will help to identify sarcopenia. Three subtests measure lower-extremity functions: keeping balance (feet side-by-side, semi-tandem, tandem balance position, to be kept for 10 seconds each), walking 4 meters at usual pace, yielding a gait speed ratio (meter per second) ; standing up and sitting down five times as quickly as possible with the arms folded. Each movement is scored 0-4 points out of a total score from 0 to 12, with higher scores showing better physical performance. If total score is under 8, there is a risk of sarcopenia. For the analyses, the variable will be dichotomized accordingly (1 = sarcopenia; 0 = no sarcopenia). The participant will complete this test at inclusion, T6 and T12.
Frailty of the participant | 12 months
  Frailty will be assessed at inclusion, T6 and T12 using Fried's phenotype (weight loss, exhaustion, low physical activity, slowness, weakness) and will be analyzed as a dichotomous variable, i.e. 1 = Fragile and 0 = Not Fragile. Information on the different components of the phenotype will be retrieved from the MNA, the SPPB and a hand-grip strength test using a dynamometer, at inclusion, T6 and T12.
Sensory impairment of the participant | 12 months
  Sensory impairments (audition and vision) will be addressed by directly asking the professional caregiver. Variables will be dichotomized accordingly ((1 = hearing / vision impairment; 0 = hearing / vision impairment). The foster caregiver will complete this questionnaire at inclusion, T6 and T12.
Activities of Daily Living of the participant | 12 months
  The level of independence in Activities of Daily Living (ADL) and incontinence will be assessed using the Katz's scale, a 6-item scale assessing independence in 6 basic activities of daily living: bathing, toileting, eating, dressing, incontinence. For each activity, a score of 1 indicates complete autonomy, a score of 0.5 indicates partial autonomy, and a score of 0 indicates complete dependency. The foster caregiver will complete this questionnaire about the participant at inclusion, T6 and T12.
Instrumental Activities of Daily Living of the participant | 12 months
  The level of independence in Instrumental Activities of Daily Living (IADL) will be assessed using Lawton's IADL scale. The foster caregiver will complete this questionnaire about the participant at inclusion, T6 and T12.
Dependency of the participant | 12 months
  In France, the AGGIR questionnaire has been developed by public authorities to quickly assess the degree of dependency of elderly people, and assign a dependency group, ranging from 0 (bedridden, completely dependent) to 6 (no help required, the person is autonomous in everyday activities.) This scale is routinely completed by every nursing home at admission and updated when necessary to reassess healthcare pathways. The foster caregiver will complete this questionnaire about the participant at inclusion, T6 and T12.
Psychological and Behavioral Symptoms in Dementia of the participant | 12 months
  Psychological and Behavioral Symptoms in Dementia will be assessed with the short version of the NeuroPsychiatric Inventory or NPI. This scale assesses presence, severity for the patient and impact on the professional's workload of an array of psychological and behavioral manifestations (agitation, hallucinations, apathy, etc.) as well as neurovegetative symptoms (sleep and appetite). The foster caregiver will complete this questionnaire about the participant at inclusion, T6 and T12.
Risk of developing pressure ulcers of the participant | 12 months
  Risk of developing pressure ulcers will be assessed with the Braden's Scale, and pressure ulcers will be classified according to the National Pressure Ulcer Advisory Panel, European Pressure Ulcer Advisory Panel and Pan Pacific Pressure Injury Alliance. The foster caregiver will complete this questionnaire about the participant at inclusion, T6 and T12.
Quality of life of the participant | 12 months
  Quality of life of the participant will be assessed using the QoL-AD (Questionnaire Quality of Life - Alzheimer's Disease). This 13-item questionnaire assesses the participant's physical condition, mood, relationships with friends and family, financial difficulties, and overall quality of life. The self-rated and the proxy-rated version of the questionnaire will be administered to the participant and the caregiver, respectively. The items are evaluated using a 4-point ordinal scale ranging from poor to excellent, with a total score ranging from 13 to 52. For the weighted score, the participant's score is multiplied by 2, the caregiver's score (about the participant's quality of life) is added, and the total is divided by 3 to bring the score back to the initial scale. The participant and the foster caregiver will complete this test at inclusion, T6 and T12.
Health-related quality of life of the participant | 12 months
  Health-related quality of life of the participant will be assessed with the EQ-5D questionnaire. This questionnaire assesses health conditions. It is the most widely used questionnaire in medico-economic analyses. It allows health outcomes to be assessed in terms of QALYs (Quality-Adjusted Life-Years). This indicator summarizes the length and quality of life in a single figure. The result of a cost-utility analysis is expressed in terms of the cost of gaining one QALY (i.e. one year lived in perfect health). To estimate QALY, health-related quality of life is designed on a continuum from 0 (death) to 1 (perfect health). Each health status is thus assigned a weight of 0 to 1, the higher the corresponding quality of life.
  The participant and the foster caregiver will complete this test at inclusion, T6 and T12
Adaptation to the foster family of the participant | 12 months
  Adaptation to the foster family will be assessed at inclusion, T6 and T12 using Castonguay & Ferron's scale. This is a 17-item scale designed to identify people who have difficulties to adjust to nursing home life, and that we adapted by replacing "nursing home" by "foster home". The participants must answer "yes" or "no" to a series of statements about their daily life and habits in the residence. A score of 16 or 17 indicates a good general adaptation, while a score of 11 or less indicates significant difficulties. The participant and the foster caregiver will complete this test at inclusion, T6 and T12
Foster caregivers' quality of life assessed with SF-36 | 12 months
  Foster caregivers' quality of life will be assessed with the Medical Outcomes Study Short-Form General Health Survey - 36 items (SF-36, a widely validated health-related quality of life questionnaire, that uses questions on physical, social and psychological domains. The foster caregiver will complete this questionnaire at inclusion and at T6 and T12.
Foster caregivers' quality of life assessed with the Pro-QoL scale | 12 months
  Symptoms of burnout will be assessed with the Pro-QoL scale (professional quality of life scale). This 30-item questionnaire yields three domain-specific scores: burnout risk, compassion, and compassion fatigue. The foster caregiver will complete this questionnaire at inclusion, T6 and T12.

CONTACTS AND LOCATIONS:
Overall Officials: Maturin MT TABUE-TEGUO, MD MhD, Principal Investigator — CHU de la Guadeloupe
Locations (1):
- University Hospital Center of Guadeloupe, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Boucaud-Maitre D, Villeneuve R, Rambhojan C, Simo-Tabue N, Thibault N, Rinaldo L, Dartigues JF, Drame M, Amieva H, Tabue-Teguo M. Clinical Characteristics of Older Adults Living in Foster Families in the French West Indies: Baseline Screening of the KArukera Study of Aging in Foster Families (KASAF) Cohort. Innov Aging. 2024 Jun 28;8(7):igae063. doi: 10.1093/geroni/igae063. eCollection 2024. PMID 39087204
- [Derived] Boucaud-Maitre D, Villeneuve R, Simo-Tabue N, Dartigues JF, Amieva H, Tabue-Teguo M. The Health Care Trajectories of Older People in Foster Families: Protocol for an Observational Study. JMIR Res Protoc. 2023 Feb 8;12:e40604. doi: 10.2196/40604. PMID 36753315